CLINICAL TRIAL: NCT01494805
Title: A Phase I/II Controlled Dose-escalating Trial to Establish the Baseline Safety and Efficacy of a Single Subretinal Injection of rAAV.sFlt-1 Into Eyes of Patients With Exudative Age-related Macular Degeneration (AMD)
Brief Title: Safety and Efficacy Study of rAAV.sFlt-1 in Patients With Exudative Age-Related Macular Degeneration
Acronym: AMD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lions Eye Institute, Perth, Western Australia (Other)
Collaborators: Adverum Biotechnologies, Inc. (Industry)
Responsible Party: Principal Investigator, Prof. P. Elizabeth Rakoczy, Principal Scientific Investigator, Lions Eye Institute, Perth, Western Australia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008-135
Record Dates: First submitted 2011-12-14; First posted 2011-12-19 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Macular Degeneration; Age-related Maculopathies; Age-related Maculopathy; Maculopathies,Age-related; Maculopathy,Age-related; Retinal Degeneration; Retinal Neovascularization; Eye Diseases
Keywords: Age-related Macular Degeneration; AAV; AMD; Wet AMD; Neovascular AMD; Gene Therapy; Ocular; Ocular Gene Therapy; Eye diseases; Macular Degeneration; Retinal Degeneration; Retinal Neovascularization; Wet Macular Degeneration; Retinal Diseases
MeSH Terms: conditions — Macular Degeneration; Retinal Degeneration; Retinal Neovascularization; Eye Diseases; Wet Macular Degeneration; Retinal Diseases | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Dose rAAV.sFlt-1 (Experimental)
  Interventions: Biological: rAAV.sFlt-1
- High Dose rAAV.sFlt-1 (Experimental)
  Interventions: Biological: rAAV.sFlt-1
- Control - ranibizumab only (Active Comparator)
  Interventions: Other: Control (ranibizumab alone)

INTERVENTIONS:
Biological: rAAV.sFlt-1 — 1 x 10^10 vector genomes (vg) rAAV.sFlt-1, delivered by subretinal injection
  Arms: Low Dose rAAV.sFlt-1
Biological: rAAV.sFlt-1 — 1 x 10^11 vector genomes (vg) rAAV.sFlt-1, delivered by subretinal injection
  Arms: High Dose rAAV.sFlt-1
Other: Control (ranibizumab alone) — Patients will not receive rAAV.sFlt-1, but will be eligible for retreatment with ranibizumab (Lucentis).
  Arms: Control - ranibizumab only

SUMMARY:
The study will involve approximately 40 subjects aged 55 or above who have exudative age-related macular degeneration (wet AMD). Patients will be randomized to receive one of two doses of rAAV.sFlt-1 or assigned to the control group.

DETAILED DESCRIPTION:
A new treatment for exudative age-related macular degeneration (wet AMD) is being investigated. The purpose of this Phase I/II clinical research study is to examine the baseline safety and efficacy of an experimental study drug to treat a complication of the disease which leads to vision loss. The name of the study drug is rAAV.sFlt-1.

This experimental study uses a non-pathogenic virus to express a therapeutic protein within the eye. The therapeutic diminishes the growth of abnormal blood vessels under the retina. The duration of effect is thought to be long-term (years) following a single administration.

The clinical research study will look at the baseline safety and efficacy of a single injection of rAAV.sFlt-1 injected directly into the eye.

Approximately forty (40) subjects will participate in Australia. The primary endpoint of the study is at one month, with extended follow up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 55 years;
* Subfoveal CNV secondary to AMD and with best corrected visual acuity of 3/60 - 6/9 with 6/60 or better in the other eye;
* Fluorescein angiogram of the study eye must show evidence of a leaking subfoveal choroidal neovascular lesion, or CNV currently under active management with anti-VEGF therapy;
* Must be a candidate for anti-VEGF intravitreal injections;
* No previous retinal treatment of photodynamic therapy or laser;
* Able to provide informed consent;
* Able to comply with protocol requirements, including follow-up visits.

Exclusion Criteria:

* Liver enzymes > 2 X upper limit of normal;
* Any prior treatment for AMD in the study / control eye, excluding anti-VEGF injections;
* Extensive sub-foveal scarring, extensive geographic atrophy, or thick subretinal blood in the study eye as determined by the investigator;
* Significant retinal disease other than sub-foveal CNV AMD;

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
No sign of unresolved ophthalmic complications, toxicity or systemic complications as measured by laboratory tests from 1 month post injection | Primary endpoint at 1 month
  1. Ocular examination:
     * Ocular inflammation
     * Intraocular pressure
     * Visual acuity
     * Retinal bleeding
  2. Abnormal laboratory data

SECONDARY OUTCOMES:
Maintenance or improvement of vision without the necessity of ranibizumab re-injections | Up to 3 years
  1. Best-corrected visual acuity
  2. CNV lesion
  3. Foveal thickness

CONTACTS AND LOCATIONS:
Overall Officials: Ian Constable, Professor, Principal Investigator — Lions Eye Institute
Locations (1):
- Lions Eye Institute, Nedlands, Western Australia, Australia

REFERENCES:
- [Derived] Constable IJ, Pierce CM, Lai CM, Magno AL, Degli-Esposti MA, French MA, McAllister IL, Butler S, Barone SB, Schwartz SD, Blumenkranz MS, Rakoczy EP. Phase 2a Randomized Clinical Trial: Safety and Post Hoc Analysis of Subretinal rAAV.sFLT-1 for Wet Age-related Macular Degeneration. EBioMedicine. 2016 Dec;14:168-175. doi: 10.1016/j.ebiom.2016.11.016. Epub 2016 Nov 10. PMID 27865764
- [Derived] Rakoczy EP, Lai CM, Magno AL, Wikstrom ME, French MA, Pierce CM, Schwartz SD, Blumenkranz MS, Chalberg TW, Degli-Esposti MA, Constable IJ. Gene therapy with recombinant adeno-associated vectors for neovascular age-related macular degeneration: 1 year follow-up of a phase 1 randomised clinical trial. Lancet. 2015 Dec 12;386(10011):2395-403. doi: 10.1016/S0140-6736(15)00345-1. Epub 2015 Sep 30. PMID 26431823